CLINICAL TRIAL: NCT04611100
Title: Efficacy of Intraductal Radiofrequency Ablation in Combination With Metallic Biliary Stenting in Advanced Hilar Cholangiocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111/2562
Record Dates: First submitted 2020-03-04; First posted 2020-11-02 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2020-03

CONDITIONS: Hilar Cholangiocarcinoma; Biliary Obstruction
Keywords: Hilar cholangiocarcinoma; Biliary obstruction; Radiofrequency ablation
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional (No Intervention): Patient receive endoscopic placement of metallic biliary stent for obstructive jaundice
- Radiofrequency ablation (Experimental): Patient receive endoscopic intraductal radiofrequency ablation before placement of biliary stent for obstructive jaundice
  Interventions: Device: ELRA endoluminal radiofrequency ablation electrode (Taewoong, Seoul, Korea)

INTERVENTIONS:
Device: ELRA endoluminal radiofrequency ablation electrode (Taewoong, Seoul, Korea) — Intraductal radiofrequency ablation using ELRA endoluminal radiofrequency ablation electrode (Taewoong, Seoul, Korea) 10W 2 minutes at the obstructed bile duct before placing uncover self-expandable biliary metal stent
  Arms: Radiofrequency ablation

SUMMARY:
The study aim to evaluate the efficacy of intraductal radiofrequency ablation for unresetable hilar cholangiocarcinoma in addition to biliary stenting. The patient would be randomized into 1:1 ratio of conventional group who received biliary stenting alone, and RFA group who receive intraductal RFA before biliary stenting. Immediate complications as well as long term stent patency and patient survival would be studied.

DETAILED DESCRIPTION:
Study design: randomized single-blind control trial Study population: patient with unresectable hilar cholangiocarcinoma with obstructive jaundice who need hilar biliary stenting Primary endpoint: Biliary stent patency time Secondary endpoint: Patient survival Intervention

1. Recruited patients randomly assigned into 2 groups, conventional and RFA group by sealed enveloped
2. All patients receive endoscopic biliary stenting. Those in RFA group receive RFA before biliary stent.
3. Monitor for adverse event during hospitalization and during follow up
4. Follow up as outpatient in 4-weekly interval with monitoring of serum liver function test as routine

ELIGIBILITY:
Inclusion Criteria:

* Hilar cholangiocarcinoma diagnosed by imaging or pathology
* Considered unresectable or unfit for surgery
* Presence of obstructive jaundice need endoscopic biliary drainage

Exclusion Criteria:

* History of unremovable metallic biliary stent placement
* severe biliary stricture that the instrument was unable to pass through
* unfit for endoscopic under conscious sedation
* loss to follow up and loss contact within 6 months after intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Biliary stent patency | up to 6 months
  The duration between primary intervention and first recurrent increased in serum total bilirubin after intervention up to 6 months after the primary procedure

SECONDARY OUTCOMES:
Patient survival | up to 6 months
  Survival time after primary intervention and documented patient death at 6 months after primary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tanyaporn Chantarojanasiri, MD, Principal Investigator — Rajavithi hospital, Bangkok, Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

REFERENCES:
- [Background] Sripa B, Pairojkul C. Cholangiocarcinoma: lessons from Thailand. Curr Opin Gastroenterol. 2008 May;24(3):349-56. doi: 10.1097/MOG.0b013e3282fbf9b3. PMID 18408464
- [Background] Doherty B, Nambudiri VE, Palmer WC. Update on the Diagnosis and Treatment of Cholangiocarcinoma. Curr Gastroenterol Rep. 2017 Jan;19(1):2. doi: 10.1007/s11894-017-0542-4. PMID 28110453
- [Background] Heimbach JK, Kulik LM, Finn RS, Sirlin CB, Abecassis MM, Roberts LR, Zhu AX, Murad MH, Marrero JA. AASLD guidelines for the treatment of hepatocellular carcinoma. Hepatology. 2018 Jan;67(1):358-380. doi: 10.1002/hep.29086. No abstract available. PMID 28130846
- [Background] Kim JH, Won HJ, Shin YM, Kim PN, Lee SG, Hwang S. Radiofrequency ablation for recurrent intrahepatic cholangiocarcinoma after curative resection. Eur J Radiol. 2011 Dec;80(3):e221-5. doi: 10.1016/j.ejrad.2010.09.019. Epub 2010 Oct 14. PMID 20950977
- [Background] Razumilava N, Gores GJ. Cholangiocarcinoma. Lancet. 2014 Jun 21;383(9935):2168-79. doi: 10.1016/S0140-6736(13)61903-0. Epub 2014 Feb 26. PMID 24581682